CLINICAL TRIAL: NCT03537092
Title: A Study of the Safety and Acceptability of a Placebo Vaginal Film: FAME101
Acronym: FAME101
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine Bunge (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Katherine Bunge, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO17090024; ES-38322 (Other: DAIDS Protocol); U19AI120249 (NIH)
Record Dates: First submitted 2018-01-16; First posted 2018-05-25 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Safety of Vaginal Film Use

STUDY DESIGN:
Intervention Model Description: All participants will insert a placebo extended release vaginal film at Day 0. They are randomized to the timing of their first follow up visit (Day 3, 7, 10 or 14) to assess how long the film can be detected visually and/or one of its components remains detectable by biochemical assay in the lower genital tract.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vaginal Film (Experimental): Each participant who inserted a single use placebo vaginal film (Day 0) is randomized to the timing of Visit 3 (Day 3, 7, 10, or 14)
  Interventions: Device: Vaginal Film

INTERVENTIONS:
Device: Vaginal Film — 2" x 2" vaginal film with no active drug

SUMMARY:
This is a phase I randomized trial assessing the safety of a single vaginal placebo film application. In order to develop a vaginal film which can provide extended release of an Antiretroviral (ARV), the film polymers and formulation have been altered from the cellulose and polyvinyl alcohol films used to deliver dapivirine and tenofovir in previous trials. Therefore, the proposed study will evaluate the safety and persistence of these film polymers when applied vaginally.

DETAILED DESCRIPTION:
This research study will involve the use of a placebo vaginal film. Investigators want to evaluate the safety of the film and understand the acceptability and length of time for the film to dissolve once inserted into the vagina. In future studies, this film may have medication added to it to deliver medication over an extended period of time (i.e. extended release).

All of the eligible women will be randomized (distributed by chance, like rolling a dice) at the Enrollment Visit to one of four study groups. The groups will specify what day Visit 3 will be performed.

Participants will have an equal likelihood of being in any one of the four groups. Neither the participant nor the study staff can choose the group or can change the group the participant has been placed into. Regardless of which group the participant is in she will only use the film once during the study. Women in all of the study groups will have the same study visit schedule except for the timing of Visit 3.

ELIGIBILITY:
Inclusion Criteria:

Women must meet all the following criteria to be eligible for inclusion in the study:

1. Age 18 through 45 years (inclusive) at screening
2. Able and willing to provide written informed consent to be screened for and to take part in the study.
3. Able and willing to provide adequate locator information
4. HIV-uninfected based on testing performed by study staff at screening (per algorithm in Appendix II)
5. In general good health as determined by the site clinician
6. Agree to be sexually abstinent for 48 hours prior to each visit and from Visit 2 to Visit 3
7. At screening, agrees to abstain from any other intravaginal product or penetration (including sex toys, excluding tampons) for 48 hours prior to each visit and between Visit 2 and 3.
8. Willingness to undergo all study-related assessments and follow all study-related procedures
9. At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products while enrolled in this trial

Exclusion Criteria:

Women who meet any of the following criteria by participant report will be excluded from the study. Of note, the study is limited to premenopausal women with an intact uterus because the mucosal immune environment differs substantially between pre- and post- menopausal women. Therefore, inclusion of post-menopausal women would introduce heterogeneity into the population.

1. Menopause (as defined as amenorrhea for one year or more without an alternative etiology)
2. Hysterectomy
3. Participant report of any of the following:

   1. Known adverse reaction to any of the study products (ever)
   2. Known adverse reaction to latex (ever)
   3. Non- therapeutic injection drug use in the 12 months prior to Screening
   4. Surgical procedure involving the pelvis in the 90 days prior to enrollment (includes dilation and curettage or evacuation, and cryosurgery; does not include cervical biopsy for evaluation of an abnormal pap smear)
   5. Participation in a drug, spermicide and/or microbicide study in the 30 days prior to enrollment or anticipated participation in an investigational drug study until completion of the study
   6. Currently pregnant or pregnancy within 42 days prior to enrollment
   7. Currently lactating
   8. Use of a diaphragm, NuvaRing®, or spermicide for contraception
   9. Internal vaginal use of any device or product (except tampons) in the 48 hours prior to enrollment
4. Urogenital infection or suspected infection within 14 days of enrollment including: symptomatic candidiasis, trichomonas vaginalis, and symptomatic bacterial vaginosis; or cervical infection, including N. gonorrhoeae, C. trachomatis, or mucopurulent cervicitis; syphilis; herpes simplex virus lesions, or other sores (Note: seropositive Herpes simplex virus without active lesions will not be excluded); acute pelvic inflammatory disease; urinary tract infection; recent exposure to a partner with N. gonorrhoeae, C. trachomatis, Trichomonas, syphilis, or nongonococcal urethritis.
5. Antibiotic or antifungal therapy (vaginal or systemic) within 7 days of enrollment
6. As determined by the PI, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease
7. Menses-like bleeding at the time of the Enrollment visit* or expected menses-like bleeding within 14 days of the Enrollment visit (*Women who have vaginal bleeding at the scheduled Enrollment Visit may return at a different date to be re-examined and possibly enrolled provided they are still within the screening window and meet all criteria.)
8. Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants must have a vagina as this is using a vaginal film
Enrollment: 64 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD, Principal Investigator — University of Pittsburgh; Sharon L Hillier, PhD, Study Chair — University of Pittsburgh
Locations (1):
- Magee womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 05/22/2018 to 11/01/2018, 84 women were recruited and screened from gynecology clinics at Magee-Womens Hospital at the University of Pittsburgh Medical Center and the surrounding community. The study was fully enrolled with 64 participants on 11/13/2018.
Period: Overall Study
Arm/Group | Vaginal Film
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vaginal Film
Number analyzed (Participants) | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26.5 [22 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic, White | 36
  Non-Hispanic, Black | 17
  Hispanic, Black | 1
  Asian | 6
  Multi-ethnic | 4
Region of Enrollment [Number; unit: participants]
  United States | 64
Marital Status [Count of Participants; unit: Participants]
  Never married | 52
  Married/domestic partner | 10
  Divorced | 1
  Separated | 1
Education [Count of Participants; unit: Participants]
  High school or less | 6
  Some college | 23
  College graduate | 27
  Trade/technical school | 8
Current smoker [Count of Participants; unit: Participants] | 13
Ever been pregnant [Count of Participants; unit: Participants] | 28
Current sexual partner [Count of Participants; unit: Participants] | 43

OUTCOME MEASURES:

1. Primary Outcome: Grade 2 or Higher Urogenital System Adverse Event Related to Film Use
Description: Any urogenital adverse event that occurs with a severity of Grade 2 (moderate) or higher that is deemed to be related to product use by the clinical primary investigator
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Film
Number analyzed (Participants) | 64
Participants | 2

2. Secondary Outcome: Correct Insertion of Vaginal Film
Description: Vaginal film was correctly inserted by the participant as assessed by clinical investigator
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Film
Number analyzed (Participants) | 64
Participants | 47

3. Secondary Outcome: Difficulty of Vaginal Film Insertion
Description: The perceived difficulty of vaginal film insertion by the participant will be assessed on a 4 point Likert scale
Time Frame: 30 days
Population: The number of participants who responded to this survey question after product insertion.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Film
Number analyzed (Participants) | 63
Participants
  Very difficult | 8
  Moderately difficult | 11
  Slightly difficult | 28
  Easy | 16

4. Secondary Outcome: Acceptability of Vaginal Film Use
Description: The acceptability of vaginal film use by the participant will be assessed on a 5 point Likert scale
Time Frame: 30 days
Population: Participants who responded to the question 'Overall I was satisfied with my experience with this film, once it was inserted' at Visit 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Film
Number analyzed (Participants) | 64
Participants
  Do not agree at all | 4
  Agree a little | 6
  Agree somewhat | 8
  Agree a lot | 20
  Agree completely | 26

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Vaginal Film
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 31/64
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Film (N=64)
Bleeding abnormality (Reproductive system and breast disorders) | 5 (5)
Genital itching (Reproductive system and breast disorders) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 7 (7)
Vaginal discharge (Reproductive system and breast disorders) | 13 (13)
Vaginal infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03537092/Prot_SAP_ICF_000.pdf